CLINICAL TRIAL: NCT05617599
Title: SUPRAFLEX CRUZPost-Market Clinical Follow-up Study
Brief Title: SUPRAFLEX CRUZ PMCF Study ( rEpic05 )
Acronym: Multiflex
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: rEpic05 - Multiflex
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: CE-MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: SUPRAFLEX CRUZ

INTERVENTIONS:
Device: SUPRAFLEX CRUZ — Patients in whom treatment with SUPRAFLEX CRUZ has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Medical Device Regulations (MDR) with multivessel coronary disease requirements in all the CONSECUTIVE patients treated with (SUPRAFLEX CRUZ).

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the SUPRAFLEX CRUZ in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old and;
* Patients treated with SUPRAFLEX CRUZ according to routine hospital practice and following instructions for use
* Patients with multivessel coronary artery disease (understood as that which affects more than one territory of the major epicardial coronary arteries - anterior descending, circumflex, right coronary artery) who is treated with more than 1 stent under study in lesions located in more than 1 of the aforementioned arteries.
* Substudy: Patients with Ejection Fraction <45% by Echocardiography
* Informed consent signed

Exclusion Criteria:

* Not meet inclusion criteria
* Contraindication for antiplatelet treatment
* Patient life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with MULTIFLEX PMCF according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Rate of target lesion failure
Device-oriented Composite Endpoint (DoCE) | 12 months
  Device-oriented Composite Endpoint (DoCE) defined as the composite of: Cardiovascular death, target vessel myocardial infarction, clinically indicated repeat revascularization of the target lesion at 12 months

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Event (MACE) | 12 months
  Composite event of cardiovascular (CV) death, non-fatal myocardial infarction (MI) and non-fatal stroke
Change from baseline in left ventricular ejection fraction (LVEF) measured by echocardiography | 1 month
  In the subgroup of patients with reduced Ejection Fraction, Change from baseline in left ventricular ejection fraction (LVEF) measured by echocardiography
Change from baseline in Global Longitudinal Strain measured by strain-rate echocardiography | 1 month
  In the subgroup of patients with reduced Ejection Fraction, Change from baseline in Global Longitudinal Strain measured by strain-rate echocardiography
Change of segmental movement of the territory revascularized measured by echocardiography | 1 month
  In the subgroup of patients with reduced Ejection Fraction, Change from baseline segmental movement of the territory revascularized measured by echocardiography
Changes in left ventricular ejection fraction (LVEF) | 1 month
  Changes in left ventricular ejection fraction (LVEF) from baseline and from 1 month post-procedure/pre-hospital discharge as assessed by echo in the subgroup of ventricular dysfunction

CONTACTS AND LOCATIONS:
Locations (21):
- Spain (21):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital General Universitario de Castellón, Castelló
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Leon, León
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Parc Tauli, Sabadell
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitario Y Politécnico La Fé, Valencia
  - Hospital Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Bangalore S, Toklu B, Patel N, Feit F, Stone GW. Newer-Generation Ultrathin Strut Drug-Eluting Stents Versus Older Second-Generation Thicker Strut Drug-Eluting Stents for Coronary Artery Disease. Circulation. 2018 Nov 13;138(20):2216-2226. doi: 10.1161/CIRCULATIONAHA.118.034456. PMID 29945934
- [Background] Lemos PA, Chandwani P, Saxena S, Ramachandran PK, Abhyankar A, Campos CM, Marchini JF, Galon MZ, Verma P, Sandhu MS, Parikh N, Bhupali A, Jain S, Prajapati J. Clinical outcomes in 995 unselected real-world patients treated with an ultrathin biodegradable polymer-coated sirolimus-eluting stent: 12-month results from the FLEX Registry. BMJ Open. 2016 Feb 17;6(2):e010028. doi: 10.1136/bmjopen-2015-010028. PMID 26888727
- [Background] Modolo R, Chichareon P, Kogame N, Asano T, Chang CC, de Winter RJ, Kaul U, Zaman A, Spitzer E, Takahashi K, Katagiri Y, Soliman OII, van Es GA, Morel MA, Onuma Y, Serruys PW. A prospective multicentre randomised all-comers trial to assess the safety and effectiveness of the thin-strut sirolimus-eluting coronary stent SUPRAFLEX: rationale and design of the Thin Strut Sirolimus-eluting Stent in All Comers Population vs Everolimus-eluting Stent (TALENT) trial. EuroIntervention. 2019 Jul 20;15(4):e362-e369. doi: 10.4244/EIJ-D-18-00499. PMID 30066672
- [Background] Zaman A, de Winter RJ, Kogame N, Chang CC, Modolo R, Spitzer E, Tonino P, Hofma S, Zurakowski A, Smits PC, Prokopczuk J, Moreno R, Choudhury A, Petrov I, Cequier A, Kukreja N, Hoye A, Iniguez A, Ungi I, Serra A, Gil RJ, Walsh S, Tonev G, Mathur A, Merkely B, Colombo A, Ijsselmuiden S, Soliman O, Kaul U, Onuma Y, Serruys PW; TALENT trial investigators. Safety and efficacy of a sirolimus-eluting coronary stent with ultra-thin strut for treatment of atherosclerotic lesions (TALENT): a prospective multicentre randomised controlled trial. Lancet. 2019 Mar 9;393(10175):987-997. doi: 10.1016/S0140-6736(18)32467-X. Epub 2019 Feb 28. PMID 30827782